CLINICAL TRIAL: NCT02921009
Title: Study of Effectiveness and Safety of Transepithelial Collagen Cross-linking at Varying Fluence Levels.
Brief Title: McNeel Eye Center Corneal Crosslinking Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McNeel Eye Center (Industry)
Responsible Party: Principal Investigator, Brian J. McNeel, O.D., F.A.A.O., McNeel Eye Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEC CxL Transepithelial
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

ARMS (1):
- Crosslinking at different fluence rates (Experimental): The study will investigate the effectiveness of Transepithelial riboflavin .25% treated with Ultraviolet light at fluence rates of 9mw/cm2 and 18mw/cm2 in the treatment of diagnosed keratoconus, pellucid marginal degeneration or post-LASIK ectasia.
  Interventions: Device: Crosslinking using UV light of two different fluence rates

INTERVENTIONS:
Device: Crosslinking using UV light of two different fluence rates — The treatment of keratoconus involves the application of riboflavin followed by Ultraviolet light of differing intensities. This study will determine the effectiveness of a greater UV light fluence at a shorter treatment time than is currently utilized.

SUMMARY:
This study will investigate the effectiveness in treating keratoconus, pellucid marginal degeneration and post LASIK iatrogenic ectasia utilizing fluence rates and treatment times of Corneal Cross Linking other than the original FDA approved protocol of 3mw/cm2.

DETAILED DESCRIPTION:
Patient recruitment will include a patient population of 100 individuals from 15 years to 50 years old with established keratoconus, pellucid marginal degeneration or post-LASIK ectasia determined by keratography. A solution of transepithelial riboflavin .25% will be applied every three minutes for 30 minutes or until complete corneal penetration is observed. Then the cornea will be irradiated with UV light at fluence rates of 9mw/cm2 for 10 minutes or 18 mw/cm2 for 5 minutes. Post procedural evaluation will take place at day one, day 7 day 30, day 90, day 180 and day 365. Pretreatment keratography, uncorrected acuity, best corrected acuity will be compared at follow up days beginning on day 30.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 15 and 50 with keratoconus diagnosed topographically with or without other corneal ectatic disease.

Exclusion Criteria:

* Prior corneal transplantation, pregnancy, inability or unwillingness to adhere to follow up protocol.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Post treatment topographic analysis of Crosslinked patients | One Year
  Pre-treatment videokeratography will be compared to post treatment keratography at certain intervals up to one year. Overall flattening of corneal curvature will be a primary study item.

SECONDARY OUTCOMES:
Post Treatment Best Corrected Visual Acuity | One Year
  Best Corrected Visual acuity will be measured post treatment out to one year. Success will be determined by improvement in best corrected acuity.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J McNeel, OD, Study Director — McNeel Eye Center; Gregory Kent, MD, Principal Investigator — The Eye Associates
Locations (1):
- McNeel Eye Center, Boise, Idaho, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with ophthalmic community once a total of 50 eyes have been completed.
Supporting Information: Study Protocol
Time Frame: Within 90 days of the completion of the study, anticipated to be in December of 2018.
Access Criteria: Via email - bjmcneelod@yahoo.com